CLINICAL TRIAL: NCT02251808
Title: Satisfaction Survey on PINS Stimulator System for Patients With Parkinson's Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Pins Medical Co., Ltd (Industry)
Collaborators: Beijing Tiantan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PINS-001
Record Dates: First submitted 2014-09-24; First posted 2014-09-29 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-05

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease, Deep brain stimulation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study will be done because the investigators would like to evaluate product satisfaction of two PINS products (product A, product B) that are to evaluate the effectiveness of rechargeable and non-rechargeable Deep Brain Stimulation (at baseline visit and at follow-up visit) and by evaluating their responses to the product satisfaction survey that will be given to them by a study coordinator.

DETAILED DESCRIPTION:
Other: IPGs products Patients implanted with the rechargeable IPGs and non-rechargeable were followed before and 3 months after DBS surgery and completed a systematic survey of satisfaction with PINS Stimulator System.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 18 to 80 years of age.
2. Subject has been diagnosed, by a neurologist, with idiopathic Parkinson's disease.
3. The PD patients can recharge the neurostimulator independently, with favourable compliance and commit to cooperate with the clinical trial study,
4. Subjects are PINS neurostimulator users

Exclusion Criteria:

Subject were major depression with suicidal thoughts (a score of >25 on the Beck Depression Inventory II,20 with scoresranging from 0 to 63 and higher scores indicating worse functioning), tumor, abnormality in routine liver and renal function, cerebral infarction, hydrocephalus, encephalatrophy, stroke sequela, heart disease, thrombocytopenia, hyperthermalgesia and any medical or psychological problem that would interfere with the conduction of the study protocol.Patients with symptoms of the midline at the state of off medication such as severe language barrier, dysphagia, disequilibrium, slipping-clutch gaitwere excluded. Patients who had undergone other implantation such as cardiac pacemaker, artificial cochlea because of the accompanied diseases such as were excluded. Patients with history of pallidotomy, stereotactic radiofrequency (Gamma Knife) and cell transplantation were also excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Of 612 patients implanted with the rechargeable IPGs and non-rechargeable (including 306 PD received rechargeable IPGs, 306 PD received non-rechargeable IPGs) were followed before and 3 months after DBS surgery and completed a systematic survey of satisfaction with PINS Stimulator System.
Sampling Method: Non-Probability Sample
Enrollment: 612 (Estimated)
Dates: Start 2014-09; Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Patient Satisfaction as Measured by Giving a Form By PINS Medical. | 3 months after DBS surgery
  Of 612 patients implanted with the rechargeable IPGs and non-rechargeable (including 306 PD received rechargeable IPGs, 306 PD received non-rechargeable IPGs) were followed before and 3 months after DBS surgery and completed a systematic survey of satisfaction with PINS Stimulator System.

CONTACTS AND LOCATIONS:
Overall Officials: Jianguo Zhang, MD, Study Director — study principal investigator
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China